CLINICAL TRIAL: NCT02484534
Title: Thrombin Generation Test in Patient With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, RAWI HAZZAN, dr, HaEmek Medical Center, Israel
Other Study IDs: EMC62-14
Record Dates: First submitted 2014-12-21; First posted 2015-06-29 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis
Keywords: Coagulation Factor; cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cirrhotic patients are patients with high morbidity and mortality, it is very important for determining the prognosis of these patients. The importance increases when these patients waiting for a liver transplant. The Model for End-Stage Liver Disease (MELD) is a reliable measure of mortality risk in patients with end-stage liver disease. It is used as a disease severity index to help prioritize allocation of organs for transplant. MELD uses the patient values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival.

Blood tests that we use today in daily practice to evaluate the coagulation system (PT, PTT) do not check actually the functioning of the system, but examine the level of clotting factors and therefore only verify that the side of Anticoagulant of the equation and not the side of the procoagulant .

To examine the coagulation system function tests have been developed, One of them is the thrombin generation. The purpose of the trial is to determine whether thrombin generation test can be a prognostic indicator in patients cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Cirrhosis patient MELD ( Model For End-Stage Liver Disease) above 12

Exclusion Criteria:

Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (men and women) who are hospitalized in internal and surgical wards with a diagnosis of cirrhosis of the liver.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2015-12-09 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Complications of cirrhosis. | 3 month.
  Complications of cirrhosis, such as ascites, bleeding Varicose veins, encephalopathy or thrombosis of the portal vein.

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek medical center, Afula, Israel